CLINICAL TRIAL: NCT00239161
Title: TREATMENT OF ACUTE UNCOMPLICATED PYELONEPHRITIS WITH SHORT COURSE LEVOFLOXACIN A Pilot Study
Brief Title: Safety and Efficacy Study of the Treatment of Kidney Infections With Short Course Levofloxacin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Ortho-McNeil Pharmaceutical (Industry); Janssen-Ortho Inc., Canada (Industry); PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPSS-353; LOF-UTI-2
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2005-10-14 (Estimated); Status verified 2005-08

CONDITIONS: Acute Uncomplicated Pyelonephritis
Keywords: Pyelonephritis
MeSH Terms: conditions — Pyelonephritis | interventions — Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin

SUMMARY:
The purpose of the study is to compare the safety and effectiveness of the antibiotic levofloxacin by administering a higher dose of levofloxacin using a shorter course of therapy to treat patients with infections of their kidney.

DETAILED DESCRIPTION:
The goal is to complete a pilot study of short course (5 days), high dose, levofloxacin treatment for women with acute uncomplicated pyelonephritis. Specific study objectives include:

1. To assess the efficacy and tolerability of levofloxacin 750 mg once daily for treatment of acute uncomplicated pyelonephritis in 25 women.
2. To describe the population pharmacokinetics of levofloxacin 750 mg once daily in treatment of young women with acute pyelonephritis.
3. To identify urine proteins associated with the inflammatory response of acute pyelonephritis, and characterize the time course of resolution of these proteins following initiation of treatment.

ELIGIBILITY:
Inclusion criteria:

* Recent onset (less than 7 days) of costovertebral angle pain or tenderness with or without fever, and with or without lower urinary tract symptoms (dysuria, frequency, urgency). Diabetic women without long term complications of diabetes (retinopathy, nephropathy, or neuropathy) may be enrolled.
* Stable hemodynamic status and able to tolerate oral medication.
* Pretherapy urine culture >107 cfu/L (>104 cfu/ml) of a uropathogen (E. coli, other Enterobacteriaceae, S. saprophyticus). Patients will be enrolled into the study prior to urine culture results being known. If pretherapy cultures are subsequently not positive (usually at 48 hours), subjects will be discontinued.
* Pyuria (> 10 wbc/mm3 or > 10 X106 wbc/L by hemocytometer; > 6-10 wbc/hpf, or > 1+ LE (leukocyte esterase) dipstick).

Exclusion Criteria:

·Pregnancy, breastfeeding, fluoroquinolone allergy, and any underlying structural or functional genitourinary abnormality.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2004-09; Study Completion 2005-07

PRIMARY OUTCOMES:
Microbiological cure at the 10-14 day and 33-35 day followup

SECONDARY OUTCOMES:
Clinical outcome at each visit. Microbiologic outcomes at 24,48,and72 hrs, adverse antimicrobial effects, adverse events or antimicrobial resistance. Correlation between pharmacodynamic parameters, bacteriologic and clinical resolution will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay E Nicolle, MD, FRCPC, Principal Investigator — University of Manitoba; Godfrey KM Harding, MD, FRCPC, Principal Investigator — University of Manitoba; George G Zhanel, PhD, FCCP, Principal Investigator — University of Manitoba
Locations (4):
- Canada (4):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba
  - Misericordia Urgent Care, Winnipeg, Manitoba
  - University of Manitoba, Winnipeg, Manitoba